CLINICAL TRIAL: NCT00000317
Title: Early Phase II Trials for Cocaine Medication Development
Brief Title: Early Phase II Trials for Cocaine Medication Development - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Research Foundation for Mental Hygiene, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: #3124; R01DA009582 (NIH); NCT00000272 (obsolete NCT alias)
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Cocaine-Related Disorders; Substance-Related Disorders
Keywords: Cocaine; METHADONE PATIENTS; RISPERIDONE
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PLacebo (Placebo Comparator): Placebo plus relapse prevention counseling
  Interventions: Drug: Placebo; Behavioral: Relapse prevention counseling
- Risperidone (Experimental): Risperidone (4mg/day) plus relapse prevention counseling
  Interventions: Drug: Risperidone; Behavioral: Relapse prevention counseling

INTERVENTIONS:
Drug: Risperidone — Risperidone (4mg/day)
  Other Names: Risperidal
  Arms: Risperidone
Drug: Placebo — Placebo
  Arms: PLacebo
Behavioral: Relapse prevention counseling — Modified manual guided relapse prevention counseling. Weekly 20 minute sessions consisting of cognitive behavioral skills. Both arms will receive this intervention.
  Other Names: RPT-CBT

SUMMARY:
The purpose of this study is to develop models for early Phase II testing of potential medications for cocaine dependence: amoxapine, risperidone and other agents.

The study was a controlled pilot trial of risperidone in opiate-dependent patients on methadone maintenance. The study explored whether risperidone reduced cocaine use, cocaine craving, and cocaine subjective effects in patients on methadone maintenance who abused cocaine and whether it had an acceptable side effect profile. This

DETAILED DESCRIPTION:
This was an 18-week prospective, randomized, placebo-controlled crossover design with placebo lead-in phase and terminal placebo phase. After two weeks of single-blind placebo, patients were randomly assigned to one of two schedules of medication:

2 Week Baseline Weeks 1-6 Weeks 7-12 Weeks 13-18 Group 1 placebo risperidone placebo placebo Group 2 placebo placebo risperidone placebo

The first 6-week phase provided an initial double-blind medication-placebo comparison. In the second six-week phase (weeks 7-12), patients crossed over to the opposite treatment. During weeks 13-18, Group 1 patients remained on placebo while Group 2 patients were tapered from risperidone to placebo. For six weeks after the end of the trial, patients were offered routine clinical treatment with counseling and psychiatrist visits as needed. Medication dosage was titrated upwards on a fixed-flexible schedule to a maximum dose of 4 mg per day. Medication began at ½ mg risperidone for 3 days, then 1 mg for four days, 2 mg per day during week 2, 3 mg per day during week 3, and 4 mg per day during weeks 4-6. The titration schedule for risperidone in weeks 7-12 was the same as for weeks 1-6. In addition to treatment as usual, patients received a modified manual-guided relapse prevention counseling program in weekly meetings lasting approximately 20 minutes; these sessions provided cognitive and behavioral skills that were found to be helpful to patients in reducing cocaine use.

ELIGIBILITY:
Inclusion:

1. good standing at methadone maintenance program
2. DSM-IV criteria for cocaine dependence or abuse
3. used cocaine at least 4 times in last month
4. able to give informed consent

Exclusion criteria

1. currently meets DSM-IV criteria for Major depression or dysthymia
2. meets DSM-IV criteria for attention deficit hyperactivity disorder, bipolar disorder, schizophrenia or any psychotic disorder
3. history of seizures
4. history of allergic reaction to risperidone
5. chronic organic mental disorder
6. significant current suicidal risk
7. pregnancy, lactation or failure to use adequate birth control (for females)
8. unstable physical disorders that may make participation hazardous
9. coronary vascular disease
10. cardiac conduction system disease as indicated by QRS duration >/= 0.11
11. current use of other prescribed psychotropic medications
12. history of failure to respond to a previous adequate trial of risperidone
13. history of neuroleptic malignant syndrome, tardive dyskinesia, or severe extrapyramidal reactions to neuroleptic medications
14. current DSM-IV criteria for another substance dependence other than nicotine.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 1996-08 (Actual); Primary Completion 1999-07 (Actual); Study Completion 1999-07 (Actual)

PRIMARY OUTCOMES:
Side effects | 1x/week for 18 weeks
  Using the Modified Systemic Assessment for Treatment Emergent Effects the psychiatrist assessed side effects
Craving | 3x/week during 18 weeks of trial
  subjective cravings were recorded on the Cocaine craving scale
Drug use | 3x/week during 18 weeks of trial
  urine drug testing and self reported use on the Substance Use Weekly Inventory
Retention | 18 weeks or length of study participation
  duration of individuals in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Nunes, M.D., Principal Investigator — NYS Psychiatric Institute
Locations (1):
- NYS Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No